CLINICAL TRIAL: NCT06126315
Title: A Randomized, Phase II/III Trial on the Biological and Clinical Effects of Acetyl-L-carnitine in ALS
Brief Title: Trial on the Biological and Clinical Effects of Acetyl-L-carnitine in ALS
Acronym: ALCALS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: University of Sydney (Other); FightMND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALCALS
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Acetylcarnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- alcar 1.5 g (Experimental): 2 pockets of ALCAR will be administered t.i.d for 48 weeks. Total daily dosage: 1.5 g
  Interventions: Drug: Acetyl-l-carnitine
- alcar 3 g (Experimental): 2 pockets of ALCAR will be administered t.i.d for 48 weeks. Total daily dosage: 3 g
  Interventions: Drug: Acetyl-l-carnitine
- placebo (Placebo Comparator): 2 pockets of placebo will be administered t.i.d for 48 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetyl-l-carnitine — Acetyl-l-carnitine
  Arms: alcar 1.5 g; alcar 3 g
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
Phase II/III multicenter, randomized, double-blind, placebo-controlled trial on acetyl-L-carnitine (ALCAR) in subjects living with amyotrophic lateral sclerosis (ALS). Primary study aim: The clinical objective consists of assessing the efficacy of ALCAR (two different dosages will be tested: 1.5g/day and 3g/day) on the progression of functional disability (loss of self-sufficiency), as measured by the ALSFRS-R scale. Secondary study aims: 1. The effect of ALCAR treatment on different clinical aspects: functional decline as measured by ALSFRS-R total score; the decline of forced vital capacity (FVC); quality of life as measured by ALSAQ-40 scale; cognitive function as measured by Edinburgh Cognitive and Behavioural ALS Screen (ECAS) scale; survival (being alive and without tracheostomy). 2. To measure the effects of ALCAR treatment on disease biomarkers potentially involved in the drug's mechanisms of action. These include PGC-1 alpha, 3-nitrotyrosine (3-NT), acetyl cyclophilin A (acetyl-PPIA), neurofilament light chain (NFL), creatine kinase (CK), Musclin/osteocrin, MyomiRNA (MiR-206), Uric acid, Matrix metalloproteinase-9 (MMP-9), Monocyte Chemoattractant Protein-1 (MCP-1), 4-Hydroxynonenal (HNE). 3. The tolerability and safety of ALCAR treatment by identifying unexpected adverse events.

Study population: 246 subjects will be enrolled on one Australian and ten Italian ALS sites.

Inclusion criteria: subjects aged 18+ years with a diagnosis of ALS according to Gold Coast Criteria; disease duration <24 months; satisfactory bulbar and spinal function (self-sufficiency evaluated by a score 3+ on the ALSFRS-R for swallowing, cutting food and handling utensils, and walking); satisfactory respiratory function (FVC ≥80% of predicted); documented progression of symptoms as measured by the ALSFRS-R scale. Disease progression rate (DFS) must be>= 0.33. DFS =(48- ALSFRS-R at screening)/months from onset to screening, treatment with Riluzole in the last four weeks. Exclusion criteria: antecedent polio infection; other motor neuron disease; involvement of other systems possibly determining a functional impairment; other severe clinical conditions; unwillingness or inability to take riluzole; previous use of ALCAR for any reason; inability to understand and comply with the study requirements, and to give written informed consent personally or via their legally authorized representative.

All eligible participants will be randomized to receive ALCAR (1,5 or 3 g/day) or placebo in addition to riluzole 50 mg b.i.d. Permuted block (with a block size of 6), 1:1:1 centralized randomization scheme will be used. The overall treatment duration will be 48 weeks. After enrolment, each participant will be followed up until death. Eligible subjects will be seen after 4, 12, 24, 36 and 48 weeks. At each visit, a general assessment will be made, including vital signs, body mass index (BMI), neurological examination (including quantitative and qualitative evaluation of the motor system), comorbidity, concomitant treatments and adverse events. Blood samples will be collected at baseline -Day 1 (randomization)-, 4, 12, 24, 36 and 48 weeks to test biomarkers. Functional disability will be assessed at each visit using the ALS-FRS-R scale. The respiratory function will be assessed using a spirometer to measure FVC before starting treatment (baseline visit) and at 4, 12, 24, 36 and 48 weeks. Cognitive function will be evaluated at baseline, weeks 24 and 48, using ECAS scale. Health-related quality of life, measured by the ALSAQ-40, will be tested at baseline, 24 and 48 weeks. Compliance will be tested by the local investigators, counting unused packages at each follow-up visit. Pre-planned statistical analyses will be done on Intention-to-treat and Per-protocol (PP) populations. The statistical plan will include descriptive statistics and a comparison of the proportions of self-sufficient participants at week 48 using the chi-square or Fisher's exact test for the primary endpoint. Secondary endpoints measured by numerical scores obtained from clinical scales will be analyzed using repeated measures mixed models, while biomarkers using repeated measures ANOVA. Time-to-event endpoints, such as survival and the probability of remaining self-sufficient over 48 weeks, will be analyzed with Kaplan-Meier curves. The number of adverse events and serious adverse events after 48 weeks will be compared between treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+;
2. ALS diagnosis according to the Gold Coast Criteria;
3. Disease duration < 24 months from symptom onset, as indicated by limb weakness or bulbar symptoms, at the randomization/baseline visit*;
4. Self-sufficiency [Satisfactory bulbar and spinal function (score 3+ on the ALSFRS-R for swallowing, cutting food and handling utensils, and walking)];
5. Satisfactory respiratory function (FVC ≥80% of predicted);
6. Documented progression of symptoms as measured by the ALSFRS-R scale. Disease progression rate (DFS) must be>= 0.33. DFS =(48- ALSFRS-R at screening)/months from onset to screening.
7. Ability to understand and comply with the study requirements;
8. Ability to give written informed consent personally or, as an alternative, via a legally authorized representative;
9. Treatment with riluzole 50 mg twice/day for at least 4 weeks prior to randomization visit;
10. Intact cognitive function, again determined by the Principal Investigator.

    * The qualifying first symptoms of ALS are limited to manifestations of weakness in extremity, bulbar, or respiratory muscles. Cramps, fasciculations, or fatigue should not be taken in isolation as a first symptom of ALS.

Exclusion Criteria:

1. Antecedent polio infection or other active infection;
2. Motor neuron disease (MND) other than ALS;
3. Involvement of other systems possibly determining a functional impairment (as measured by the endpoints) for the entire duration of the study;
4. Other severe clinical conditions (e.g., cardiovascular disorders, neoplasms) with an impact on survival or functional disability in the next 12 months;
5. Previous use of ALCAR for any reason;
6. Poor compliance with previous treatments;
7. Other experimental treatments in the three months prior to the screening visit (if a subject is receiving another experimental drug, a 3-month wash-out period before participating in the present clinical trial will be required);
8. Women who are lactating or able to become pregnant (e.g. who are not post-menopausal, surgically sterile, or using inadequate birth control) and men unable to practice contraception for the duration of the treatment and three months after its completion;
9. Inability to understand and comply with the study requirements;
10. Unwillingness or inability to take riluzole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
self-sufficient | 48 weeks
  The proportion of participants remaining self-sufficient after 48 weeks in each treatment arm

SECONDARY OUTCOMES:
Mean change of ALSFRS-R total score in each treatment arm | from baseline to week 48
  Mean change of ALSFRS-R total score in each treatment arm
Mean change of FVC% in each treatment arm | from baseline to week 48
  Mean change of FVC% in each treatment arm
Mean change in the five domains of ALSAQ-40 measuring different aspects of quality of life (physical mobility, ADL/independence, eating and drinking, emotional reactions, communication) in each treatment arm | from baseline to week 48
  Mean change in the five domains of ALSAQ-40 measuring different aspects of quality of life (physical mobility, ADL/independence, eating and drinking, emotional reactions, communication) in each treatment arm
Mean change in ECAS total score in each treatment arm | from baseline to week 48
  Mean change in ECAS total score in each treatment arm
Cumulative probability of remaining self-sufficient in each treatment arm | from baseline to week 48
  Cumulative probability of remaining self-sufficient in each treatment arm
Cumulative probability of remaining free from a 6-point or greater decline in ALSFRS-R total score in each treatment arm | from baseline to week 48
  Cumulative probability of remaining free from a 6-point or greater decline in ALSFRS-R total score in each treatment arm
Cumulative probability of remaining without gastrostomy in each treatment arm | from baseline to week 48
  Cumulative probability of remaining without gastrostomy in each treatment arm
Cumulative probability of remaining without non-invasive ventilation (NIV) support (≥12 hours a day in a 24-hour period) in each treatment arm | from baseline to week 48
  Cumulative probability of remaining without non-invasive ventilation (NIV) support (≥12 hours a day in a 24-hour period) in each treatment arm
Cumulative survival probability (of being alive and without tracheostomy) in each treatment arm | from baseline to week 48
  Cumulative survival probability (of being alive and without tracheostomy) in each treatment arm
The mean change in the levels of PGC-1 alpha, 3-NT, acetyl-PPIA in the peripheral blood mononuclear cells (PBMCs) and of NFL, MMP-9, MCP-1, CK, MiR-206, Musclin/osteocrin, Uric acid, HNE in plasma in each treatment arm, during the entire treatment period | from baseline to week 48
  The mean change in the levels of PGC-1 alpha, 3-NT, acetyl-PPIA in the peripheral blood mononuclear cells (PBMCs) and of NFL, MMP-9, MCP-1, CK, MiR-206, Musclin/osteocrin, Uric acid, HNE in plasma in each treatment arm, during the entire treatment period
Number of adverse events and serious adverse events in each treatment arm | from baseline to week 48
  Number of adverse events and serious adverse events in each treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Pupillo, PharmD, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (19):
- Concord Hospital, Sydney, Australia
- Italy (18):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Dipartimento di Neurologia, Bergamo
  - Fondazione Serena ONLUS Centro Clinico NEMO Brescia, Brescia
  - Istituto Auxologico Italiano, IRCCS Dipartimento di Neurologia, Milan
  - Fondazione Serena ONLUS centro clinico NEMO, Milan
  - AOU di Modena Nuovo Ospedale Civile S. Agostino Estense di Modena - Ospedale di Baggiovara, Modena
  - Azienda Ospedaliera Universitaria Federico II Di Napoli, Napoli
  - Azienda Ospedaliera Universitaria "Luigi Vanvitelli", Dipartimento di Scienze mediche e chirurgiche avanzate, Napoli
  - Azienda Ospedaliero-Universitaria Maggiore della Carità, Novara
  - Azienda Ospedale-Università di Padova, Unità di Neurologia Clinica, Padua
  - A.S.P. Palermo, Villa delle Ginestre Hospital, Palermo
  - Fondazione Mondino Istituto Neurologico Nazionale a Carattere Scientifico IRCCS, Pavia
  - Fondazione Serena ONLUS-Centro Clinico NEMO Trento, Pergine Valsugana
  - Azienda Ospedaliera di Perugia, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliero Universitaria Pisana, Dipartimento di Medicina Clinica e Sperimentale, Pisa
  - San Camillo Forlanini Hospital, Center for Neuromuscolar and Neurological Rare Diseases, Unit of Neurology and Neurophysiopathology, Roma
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I - Università di Roma "La Sapienza", Roma
  - Fondazione Serena ONLUS - Centro Clinico NeMO Ancona, Torrette

IPD SHARING:
Plan to Share IPD: No